CLINICAL TRIAL: NCT07027072
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Finding, Phase 2a Clinical Trial to Evaluate the Efficacy and Safety of KDS2010 in Patients With Alzheimer's Disease With Mild Cognitive Impairment and Mild Dementia Due to Alzheimer's Disease
Brief Title: Study to Evaluate the Efficacy and Safety of KDS2010 in Patients With Alzheimer's Disease With Mild Cognitive Impairment and Mild Dementia Due to Alzheimer's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroBiogen Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NB_KDS_ADP2_23; KCT0010589 (Registry Identifier: CRIS)
Record Dates: First submitted 2025-05-15; First posted 2025-06-18 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment (MCI); Mild Dementia; Alzheimer's Disease
Keywords: Mild Cognitive Impairment; Mild Dementia; KDS2010; MAO-B inhibitor; Alzheimer's Disease
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled, Dose-Finding, Phase 2a Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A double-blind design is used to ensure scientific validity. Subjects and investigators are unaware of treatment allocation, with identical appearance between the drug and placebo. Randomization numbers are used for subject identification, and group assignments are disclosed only after the end of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group_Placebo (Placebo Comparator): A placebo will be administered orally once daily as two tablets per day for 24 weeks. This group will match the investigational drug in appearance but contain no active ingredients to maintain blinding.
  Interventions: Drug: Placebo
- Treatment Group 1_KDS2010 60 mg (Experimental): KDS2010 60 mg will be administered orally once daily as two tablets per day (one 60 mg KDS2010 tablet and one placebo tablet, 60 mg total) for 24 weeks. This group will receive the active investigational drug to evaluate its safety and efficacy.
  Interventions: Drug: KDS2010
- Treatment Group 2_KDS2010 120 mg (Experimental): KDS2010 60 mg will be administered orally once daily as two tablets per day (two 60 mg KDS2010 tablets, 120 mg total) for 24 weeks. This group will receive the higher dose of the investigational drug to evaluate its safety and efficacy.
  Interventions: Drug: KDS2010

INTERVENTIONS:
Drug: KDS2010 — KDS2010 will be administered orally once daily, two tablets per day, for 24 weeks. Dosage will be either 60 mg or 120 mg depending on the assigned group.
  Arms: Treatment Group 1_KDS2010 60 mg; Treatment Group 2_KDS2010 120 mg
Drug: Placebo — Placebo matching the investigational product in appearance but containing no active ingredient, administered orally once daily, two tablets per day, for 24 weeks.
  Arms: Control Group_Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, dose-finding Phase 2a clinical trial will be conducted to evaluate the efficacy and safety of KDS2010 in patients with Mild Cognitive Impairment (MCI) due to Alzheimer's disease (AD) and mild dementia due to Alzheimer's disease.

Based on preliminary efficacy observed in the Phase 1 clinical trial, a multinational study will be conducted in both Korea and the United States. Eligible patients diagnosed with MCI or mild Alzheimer's disease will be stratified by disease stage (MCI/mild AD) and geographic region (Korea/USA) prior to randomization. Subjects will be randomly assigned in a 1:1:1 ratio to either Treatment Group 1, Treatment Group 2, or the Control Group. The investigational product will be administered orally once daily for a duration of 24 weeks. Approximately 114 subjects will be enrolled, including an estimated 20% dropout rate, with 38 subjects assigned to each group (Treatment Group 1, Treatment Group 2, and Control Group).

The objectives of the study are as follows:

1. Efficacy Objectives: Efficacy will be evaluated through changes in cognitive function, self-management, and daily living activities before and after administration of KDS2010. Biomarker analysis in plasma and in cerebrospinal fluid (CSF; optional) will also be conducted to explore treatment efficacy.
2. Safety Objectives: The safety and tolerability will be evaluated after administration of KDS2010.
3. Exploratory Objectives: The efficacy of Treatment Groups 1 and 2 compared to the Control group will be explored through cognitive endpoints (the Clinical Dementia Rating-Sum of Boxes (CDR-SB), the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog13), and the Mini-Mental State Examination (MMSE)), stratified by demographic information, tauopathy, and ApoE4 genes.

Based on nonclinical and Phase 1 clinical data, KDS2010 will be administered orally once daily at two dose levels: 60 mg and 120 mg.

DETAILED DESCRIPTION:
This Phase 2a, multinational, randomized, double-blind, placebo-controlled, dose-finding clinical trial is designed to evaluate the efficacy, safety, and pharmacokinetics of KDS2010, a novel investigational product, reversible monoamine oxidase-B (MAO-B) inhibitor, in patients with Alzheimer's Disease (AD) with Mild Cognitive Impairment (MCI) and Mild Dementia due to Alzheimer's Disease. The clinical trial is conducted at selected sites in Korea and the United States.

A total of 114 subjects are planned for the study, with 38 subjects in each of the three groups: two treatment groups (receiving different doses of KDS2010) and a placebo control group. Subjects will be randomized in a 1:1:1 ratio, and the study is designed to allow for a 20% dropout rate. Inclusion criteria require that participants be aged between 50 and 85 years, diagnosed with MCI or mild AD, and amyloid-positive as confirmed by PET scans. Eligible participants must also demonstrate cognitive impairment as indicated by a CDR score between 0.5 and 1.0 and an MMSE score between 21 and 30.

Key exclusion criteria include individuals with cognitive impairment caused by conditions other than AD, those with a history of serious medical conditions such as cardiovascular disease or cancer, and individuals who have used AD-modifying agents or CNS-active drugs within 12 weeks prior to screening.

The primary efficacy endpoint is the change in cognitive function, assessed through the Clinical Dementia Rating-Sum of Boxes (CDR-SB), Mini-Mental State Examination (MMSE), and Alzheimer's Disease Assessment Scale-Cognitive 13 (ADAS-Cog13) scores. Secondary efficacy endpoints include changes in daily living activities (measured by the Activities of Daily Living Scale and the Alzheimer's Disease IADL Questionnaire), as well as biomarkers such as tauopathy and Apo-E4. Exploratory endpoints will assess cognitive decline and specific changes in brain imaging (e.g., PET scans) and cerebrospinal fluid biomarkers.

Safety will be evaluated through monitoring adverse events (AEs), vital signs, laboratory tests, ECGs, and psychological assessments, including the Columbia-Suicide Severity Rating Scale (C-SSRS). Pharmacokinetic parameters (AUCtau, Cmax,ss, Cmin,ss, Cav,ss, Tmax,ss, T1/2, and PTF, etc.) will be measured to assess systemic exposure to KDS2010.

Subjects must be aged between 50 and 85 years, diagnosed with MCI or mild AD, and amyloid-positive based on PET scan results. Inclusion criteria also require cognitive impairment as indicated by a CDR score between 0.5 and 1.0 and an MMSE score between 21 and 30. Major exclusion criteria include conditions other than AD that cause cognitive impairment, uncontrolled systemic diseases, and recent use of AD-modifying agents.

The primary aim of the study is to determine the potential of KDS2010 to slow cognitive decline in individuals with early-stage Alzheimer's disease, with secondary and exploratory objectives focused on safety, quality of life, and understanding the drug's pharmacokinetic profile. This study aims to provide important insights into the potential therapeutic benefits of KDS2010 in treating Alzheimer's disease at the early stages of cognitive decline.

The total duration of the study is expected to be approximately 30 months from IRB/IEC approval, with individual subject participation lasting up to 9 months. This trial aims to evaluate the safety, efficacy, and pharmacokinetics of KDS2010 as a potential treatment for early stages of Alzheimer's disease, with the goal of advancing the development of KDS2010 in the treatment of AD.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged ≥50 and ≤85 years at the time of written consent
* Patients with MCI or mild AD confirmed at screening according to the 2024 diagnostic criteria (APPENDIX 1) of the National Institute on Aging-Alzheimer's Association (NIA-AA)
* Subjects whose total CDR score (CDR-GS) is 0.5 to 1.0 at screening (however, CDR memory score is ≥0.5)
* Subjects with a Mini-Mental State Examination (MMSE) score of 21 to 30 at screening
* Subjects who test positive for amyloid on Positron Emission Tomography (PET) during screening
* Subjects who have a caregiver capable of providing accurate information about the subject's cognitive and functional abilities and appropriate for the planned assessments in the study, as judged by the investigator
* Subjects (or their legal representatives) who have voluntarily agreed to participate in this study and have given written consent

Exclusion Criteria:

* Cognitive impairment or dementia due to causes other than Alzheimer's disease

  * Vascular dementia, central nervous system infections (e.g., HIV, syphilis, etc.), head trauma, Creutzfeldt-Jakob disease, Pick's disease, Huntington's disease, Parkinson's disease, subdural hematoma, normal pressure hydrocephalus, brain tumor, thyroid disorders, parathyroid disorders, Vitamin B12 deficiency, folic acid deficiency, other metabolic and nutritional deficiencies, etc.
  * Alcohol or drug abuse, dependence
* Subjects with cognitive impairment due to hypothyroidism, nutritional deficiencies, Vitamin B12 or folic acid deficiency as assessed during screening
* Subjects confirmed during screening to have had the following medical history:

  * Malignant tumors within five years prior to screening except for basal cell carcinoma, cutaneous squamous cell carcinoma, thyroid cancer, or carcinoma in situ that has not recurred in over three years and is considered successfully treated by the investigator
  * History of alcohol or drug abuse within two years prior to screening
  * Loss of consciousness of unknown cause, or seizure within the past 52 weeks before screening
  * Unstable and clinically significant cardiovascular diseases despite appropriate treatment (acute coronary syndrome (ACS), tachycardia, clinically significant arrhythmias, cardiomyopathy, angina of at least CSS III, heart failure of NYHA II-IV, or clinically significant valvular heart disease) within 24 weeks before baseline
  * Severe or active infectious diseases requiring antibiotics or antivirals within four weeks before baseline
  * A history of stroke involving a major vascular area, transient ischemic attack (TIA), epilepsy, or severe head trauma with loss of consciousness
  * Hypersensitivity or allergy to any components of the investigational product
* Subjects confirmed during screening to have had the following accompanying disease:

  * Clinically significant neurological diseases or serious pathological findings affecting cognitive function as confirmed by brain imaging studies within 52 weeks prior to screening, including multiple sclerosis, normal pressure hydrocephalus, brain tumor (however, exceptions are allowed for lesions diagnosed as benign and with a maximum diameter of less than 1 cm), spinal cord infarction, major hemorrhage (defined as having a diameter > 1 cm in MRI) or subdural hemorrhage, cerebral vascular malformation, communicating hydrocephalus, inflammatory demyelinating diseases, etc.
  * Uncontrolled hypertension despite appropriate treatment at screening or baseline (SBP ≥160 mmHg or DBP ≥100 mmHg)
  * Dizziness or fainting when standing due to orthostatic hypotension that may affect the evaluation according to the judgment of the investigator
  * Uncontrolled diabetes (HbA1c > 9%) during screening, despite appropriate treatment
  * Bleeding disorders (Platelet <50,000/mm³) during screening, despite appropriate treatment
  * Patients with severe hepatic impairment (Child-pugh class C) at screening
  * Following laboratory test values at screening:

    * AST or ALT > 2.5 x ULN
    * total bilirubin > 1.5 x ULN (however, in case of Gilbert syndrome, > 3.0 mg/dL)
    * MDRD eGFR < 30 mL/min/1.73 m²
  * QTcF interval >450 msecs (12-lead ECG) during screening
  * Gastrointestinal diseases that may affect oral administration or absorption (celiac disease, Crohn's disease, intestinal resection, etc.)
  * Gastrointestinal diseases, including gastric and duodenal ulcers, that may affect the safety evaluation according to the judgment of the investigator
  * Psychiatric diagnosis or symptoms that may interfere with the study (uncontrolled major depression, uncontrolled schizophrenia, uncontrolled bipolar affective disorder, etc.), as assessed by the investigator
  * Positive responses to items 4 or 5 on the Columbia University Suicide Severity Rating Scale (C-SSRS) during screening
  * Other conditions deemed by the investigator to potentially affect the outcome of the study
* Subjects who have undergone or require treatment with the following:

  * AD disease-modifying agents (aducanumab, lecanemab, donanemab, gantenerumab, solanezumab, blarcamesine, simufilam, tricaprilin, valiltramiprosate, etc.) within 12 weeks before screening
  * Medications that may improve cognitive abilities or affect AD treatment (AChEIs, donepezil, galantamine, rivastigmine, tacrine, memantine, etc.) within 12 weeks before screening, except if the subject has been on a stable dose for at least 12 weeks before baseline and maintains the same composition/dosage/method of administration during the study period
  * CNS-active drugs or those affecting cognitive function antidepressants other than serotonergic drugs [e.g., bupropion], sedatives [e.g., carbamazepine], dopamine antagonists [e.g., antipsychotics, metoclopramide], amfepramone, mazindol) within 12 weeks before screening
  * Central anticholinergics and sedating H1-antihistamines within 12 weeks before screening.

However, exceptions are allowed for one-time use of the drugs, such as second-generation H1 antihistamines (e.g., cetirizine, levocetirizine, etc.) or peripheral anticholinergics with no central action (e.g., trospium for treating overactive bladder). But the use is prohibited for at least 3 days from the date of cognitive function evaluation.

* Other investigational products or clinical trial devices within four weeks before baseline or five times the half-life of the drug (whichever is longer, and patients can be enrolled after wash-out)
* Monoamine oxidase inhibitors (MAOIs) and linezolid within two weeks before baseline or five times the half-life of the drug (whichever is longer, and patients can be enrolled after wash-out)
* Opioids (pethidine, tramadol, tapentadol, etc.) within two weeks before baseline or five times the half-life of the drug (whichever is longer, and patients can be enrolled after wash-out)
* Cyclobenzaprine and St. John's wort within two weeks before baseline or five times the half-life of the drug (whichever is longer, and patients can be enrolled after wash-out)
* The following serotonergic drugs within two weeks before baseline or five times the half-life of the drug (whichever is longer, and patients can be enrolled after wash-out),

  * selective serotonin (5HT1) agonists
  * lithium
  * lamotrigine
  * ritonavir
  * dapoxetine
  * Selective serotonin reuptake inhibitors (SSRIs)
  * dapoxetine
  * Serotonin-norepinephrine reuptake inhibitors (SNRIs)
  * Tricyclic or tetracyclic antidepressants
  * triazolopyridine antidepressant However, amitriptyline ≤ 50 mg/day, trazodone ≤ 100 mg/day, citalopram ≤ 20 mg/day, and sertraline ≤ 100 mg/day are allowed without washout.
* Use of sympathomimetics (ephedrine, methylphenidate, amphetamine, methamphetamine, lisdexamfetamine, etc.) during the screening period
* Use of Dextromethorphan during the screening period
* Use of CYP3A4 strong inducer, CYP3A4 strong inhibitor, CYP2D6 strong inducer, and CYP2D6 strong inhibitor during the screening period

  * Inability to undergo MRI or PET scans
  * Pregnant or breastfeeding women
  * Fertile women or men who are unwilling to use effective contraception* from the date of written consent until 12 weeks after the last administration of the investigational product

    *Effective contraception is defined as follows, and at least one method should be used:
    * Hormonal contraception (oral, injectable, implantable, etc.)
    * Intrauterine device (IUD) or system (IUS)
    * Sterilization or surgical procedures (vasectomy, bilateral tubal ligation/surgery, hysterectomy)
    * Dual contraception methods: Simultaneous use of barrier methods (male condoms) with the methods listed above
    * Absolute abstinence: Total abstinence from sexual intercourse is recognized if the investigator deems the subject's age, occupation, lifestyle, or sexual orientation assures contraception. However, periodic abstinence (calendar method, mucus method, and symptothermal method), withdrawal, and coitus interruptus are not recognized as effective contraception methods.
  * Other conditions deemed by the investigator to be unsuitable for participation in the study

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Clinical Dementia Rating - Sum of Boxes (CDR-SB) score | Screening (-8 Week~), Week 4, Week 8, Week 12, Week 24, Week 26
  Clinical Dementia Rating (CDR) is a tool developed to assess the clinical stages of Alzheimer's disease. CDR 0 indicates "no dementia," CDR 0.5 "questionable," CDR 1 "mild," CDR 2 "moderate," and CDR 3 "severe" dementia. The range for CDR-SB is 0 to 18 points, where higher scores indicate more severe dementia.
Time to ≥0.5-point increase in CDR-SB | Up to Week 26
  Time from randomization to the first occurrence of ≥0.5-point increase in CDR-SB score.
Change from Baseline in Mini-Mental State Examination (MMSE) score | Screening (-8 Week~), Week 12, Week 24, Week 26
  The MMSE is a cognitive function and disease severity assessment composed of 30 items. Each is graded on a 2-point scale where 1 point is awarded for correct performance and 0 points if not performed correctly. Lower total scores on the MMSE indicate cognitive impairment.
Change from Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog13) score | Screening (-8 Week~), Week 12, Week 24, Week 26
  ADAS-Cog13 is a comprehensive tool for the early diagnosis of dementia and the sensitive assessment of disease progression stages. The assessment includes 9 "neuropsychological tests" and 4 "clinical assessments of cognitive damage", totaling 13 items. The higher the total score of the ADAS-Cog, the more it indicates cognitive dysfunction.
Change from Baseline in Amsterdam Instrumental Activities of Daily Living Questionnaire (A-IADL-Q-SV) score | Screening (-8 Week~), Week 12, Week 24
  The A-IADL-Q is a questionnaire designed to assess impairments in instrumental activities of daily living (IADL) in patients with dementia. The A-IADL-Q-SV is a short version of the A-IADL-Q, consisting of 30 items that assess instrumental daily functioning sensitive to cognitive decline. Each item is rated on a 5-point Likert scale, with higher scores indicating better functional ability.

SECONDARY OUTCOMES:
Percentage change from Baseline in plasma and Cerebrospinal Fluid(CSF) biomarkers | Screening (-8 Week~), Week 12, Week 24
  Changes in plasma and CSF levels of MAO-B (Monoamine Oxidase B) specific activity, GFAP (Glial Fibrillary Acidic Protein), P-tau181 (Phosphorylated-Tau 181), P-tau217 (Phosphorylated-Tau 217), Aβ-40 (Amyloid beta 40), Aβ-42 (Amyloid beta 42), NfL (Neurofilament Light Chain), BDNF (Brain-derived Neurotrophic Factor), IL-1β (Interleukin-1β), and TNF-α (Tumor Necrosis Factor-α).
Percentage change from Baseline in plasma Monoamine Oxidase B (MAO-B) specific activity | Screening (-8 Week~), Week 26
  Plasma MAO-B specific activity at Week 26 compared to baseline.

OTHER OUTCOMES:
Number of subjects with treatment-related Adverse Events (AEs) | Through study completion (approx. 26 weeks)
  AEs will be coded using MedDRA and assessed for severity and causality using CTCAE v5.0. The number of subjects affected and the incidence rates will be presented for each treatment group.
Change from baseline in systolic and diastolic blood pressure | Screening (-8 Week~), Baseline (Week 0), Week 4, Week 8, Week 12, Week 24, Week 26
  Blood pressure will be measured in mmHg at each visit.
Change from baseline in pulse rate | Screening (-8 Week~), Baseline (Week 0), Week 4, Week 8, Week 12, Week 24, Week 26
  Pulse rate will be measured in beats per minute.
Change from baseline in body temperature | Screening (-8 Week~), Baseline (Week 0), Week 4, Week 8, Week 12, Week 24, Week 26
  Body temperature will be measured using a standard thermometer.
Change from baseline in laboratory test results | Screening (-8 Week~), Baseline (Week 0), Week 4, Week 8, Week 12, Week 24, Week 26
  Laboratory parameters, including routine hematology, blood chemistry, coagulation, urinalysis, and others, will be measured. Change from baseline will be analyzed.
Change from baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) total score | Screening (-8 Week~), Week 24
  C-SSRS is used to assess the risk of suicide through interviews with the subject. The scores of each question are summed to range from 0 to 25 points. If "yes" from questions 4 or 5, categorize a subject as high-risk, requiring further evaluation, while other scores indicate a lower risk.
Pharmacokinetic Parameters: Area Under the Plasma Concentration-Time Curve over the dosing interval (τ) (AUCtau) at steady-state | Baseline (Week 0), Week 12
  AUCtau is the area under the plasma concentration-time curve over the dosing interval (τ) at steady-state, and it reflects the extent of drug exposure within a dosing cycle.
Pharmacokinetic Parameters: Peak Plasma Concentration at Steady State (Cmax,ss) | Baseline (Week 0), Week 12
  The highest plasma drug concentration observed during a dosing interval at steady state.
Pharmacokinetic Parameters: Minimum Plasma Concentration at Steady State (Cmin,ss) | Baseline (Week 0), Week 12
  The lowest plasma drug concentration during a dosing interval at steady state, usually occurring right before the next dose.
Pharmacokinetic Parameters: Average Plasma Concentration at Steady State (Cav,ss) | Baseline (Week 0), Week 12
  The average plasma concentration over the dosing interval at steady state. Calculated as: Cav, ss = AUCtau/τ
Pharmacokinetic Parameters: Time to Maximum Plasma Concentration at Steady State (Tmax,ss) | Baseline (Week 0), Week 12
  The time taken to reach the maximum plasma concentration after dosing at steady state.
Pharmacokinetic Parameters: Terminal Elimination Half-life (t1/2) | Baseline (Week 0), Week 12
  The time required for the plasma concentration of the drug to decrease by half.
Pharmacokinetic Parameters: Peak-Trough Fluctuation at Steady State (PTF) | Baseline (Week 0), Week 12
  A measure of the fluctuation between the peak (Cmax,ss) and trough (Cmin,ss) plasma concentrations during a dosing interval.

CONTACTS AND LOCATIONS:
Overall Officials: Sangwook Kim, Chief Executive Officer, Study Director — NeuroBiogen Co., Ltd
Locations (8):
- South Korea (8):
  - Chonnam National Unversity Hospital, Gwangju, Gwangju
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - The Catholic University of Korea St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon, Incheon
  - Hanyang University Seoul Hospital, Seoul, Seoul
  - Konkuk University Medical Center, Seoul, Seoul
  - Asan Medical Center, Seoul, Seoul

IPD SHARING:
Plan to Share IPD: No